CLINICAL TRIAL: NCT07211880
Title: A Community-based Collaborative Study for Eradication of Helicobacter Pylori and Associated Gastric Cancer in Bhutan
Brief Title: Helicobacter Pylori Infection and Gastric Disease in Bhutan: First Community-Wide, Population-Based Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zero Helicobacter IGAN Network (Other)
Collaborators: Oita University (Other); Japan International Cooperation Agency (Other); JDWNRH (Other); Khesar Gyalpo University of Medical Sciences of Bhutan (Unknown); Royal Centre for Disease Control Bhutan (Unknown)
Responsible Party: Principal Investigator, Yumiko Kamogawa, M.D., Ph.D. President of Zero Helicobacter IGAN Network, Zero Helicobacter IGAN Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO/2019/076
Record Dates: First submitted 2025-09-19; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: H.Pylori; Gastric Cancer; H Pylori Eradication
Keywords: H. pylori; gastric cancer; H pylori eradication triple therapy; Bhutan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Rabeprazole; Clarithromycin; Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: Screening of H pylori and eradication in order to prevent gastric cancer using community-based longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H pylori positive individual (Experimental): H pylori positive individual receiving triple therapy
  Interventions: Drug: Rabeprazole Sodium, Amoxicillin Hydrate, Clarithromycin; Diagnostic Test: Upper gastrointestinal endoscopy for the H. pylori and serum pepsinogen positive individuals (high risk group of gastric cancer)
- H. pylori positive individuals for UBT test (Experimental): The H pylori positive individuals are treated by triple therapy. After 6-8 weeks, the eradication is confirmed by using the UBT (13C Urea Breath Test: Beijing Richen-force Science & Technology Co. Ltd).
  Interventions: Device: Urea Breath Test for the prevalence of H pylori

INTERVENTIONS:
Drug: Rabeprazole Sodium, Amoxicillin Hydrate, Clarithromycin — 7 days therapy
  Arms: H pylori positive individual
Diagnostic Test: Upper gastrointestinal endoscopy for the H. pylori and serum pepsinogen positive individuals (high risk group of gastric cancer) — Endoscopic examinations were conducted using a GIF-150 endoscope in combination with the CV150 system (Olympus Co., Tokyo, Japan).
  Arms: H pylori positive individual
Device: Urea Breath Test for the prevalence of H pylori — After eradication of the H pylori with drug success of the therapy was assessed 6 to 8 weeks after treatment using the UBT(C13 Urea Breath Test: Beijing Richen-Force Science & Techinology Co. Ltd.)
  Arms: H. pylori positive individuals for UBT test

SUMMARY:
Background: Helicobacter pylori is a major risk factor for gastric cancer, yet in many developing countries, including Bhutan where gastric cancer incidence is high, access to screening and eradication is limited. The investigators conducted the first large-scale, population-based survey of H. pylori infection and gastric disease in Bhutan to provide baseline data before the launch of a national gastric cancer prevention program.

Methods: Permanent residents aged ≥12 years from 24 villages under Dawakha Basic Health Unit II catchment area were enrolled (December 2019-March 2023). H. pylori status was determined by serum IgG testing, gastric atrophy by serum pepsinogen, and endoscopy was offered to high-risk groups.

DETAILED DESCRIPTION:
The investigators enrolled permanent residents aged ≥12 years living in communities within the catchment area of Dawakha BHU II, Paro District, Bhutan, between December 2019 and March 2023. The objectives of this study were to evaluate the status of H. pylori infection, the prevalence of endoscopic gastric diseases including gastric cancer and peptic ulcers, and to provide eradication therapy for infected individuals. Exclusion criteria included individuals with medical conditions in which triple therapy or endoscopy was contraindicated (e.g., pregnancy, renal disease, history of respiratory difficulty), those with a prior history of H. pylori eradication therapy, and individuals who declined to provide informed consent.

The study protocol complied with the ethical principles of the Declaration of Helsinki and was approved by the Institutional Review Board of Khesar Gyalpo University of Medical Sciences of Bhutan (approval number: PO/2019/076). Written informed consent was obtained from all participants. This prospective clinical trial was registered on July 1, 2021, in the University Hospital Medical Information Network (UMIN), under the identifier UMIN000044707 (http://www.umin.ac.jp/ctr/index.htm).

All participants underwent H. pylori serological testing and measurement of serum pepsinogen levels to assess infection status and evaluate the degree of serological gastric atrophy, respectively.

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female age 12 years and above in the selected communities for H. pylori infection screening

  * Both male and female age 18 years and above in the selected communities for H. pylori infection screening, eradication and endoscopy.
  * Permanent residence of the communities

Exclusion Criteria:

* Exclusion criteria for screening

  * Individuals not consenting Exclusion criteria for eradication and endoscopy
  * Pre-existing medical conditions where triple therapy or endoscopy is not recommended (mainly pregnant women, renal diseases, history of breathing difficulty)

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1043 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of H. pylori | 2 months
  The seroprevalence of H. pylori (IgG ≥10 U/m) as positive for the H pylori
Gastric atrophy by pepsinogen test | 2 Months
  As a marker of gastric atrophy, serum levels of pepsinogen I and II were measured using a chemiluminescence enzyme immunoassay (E-Plate Eiken Disc Pepsinogen I and II; Eiken Chemical Co., Ltd., Tochigi, Japan). A positive result in the pepsinogen method was defined as a pepsinogen I level ≤70 ng/mL and a pepsinogen I/II ratio ≤3. Based on the results of both the pepsinogen test and H. pylori IgG levels, participants were classified into four ABC groups (A-D), which reflect the risk of gastric cancer according to the ABC method.

SECONDARY OUTCOMES:
Gastrointestinal endoscopic examination | 3 months
  Based on the results of the serological tests, upper gastrointestinal endoscopy was performed in participants classified as ABC group, C or D( as high risk of gastric cancer group), as well as those classified as group B who were over 40 years of age. In addition, endoscopy was also conducted for individuals who voluntarily requested the procedure, regardless of their ABC classification.
H pylori eradication therapy | 3 months
  Patients diagnosed with H. pylori infection received a standard 7-day triple therapy regimen consisting of rabeprazole (10 mg twice daily), amoxicillin (750 mg twice daily), and clarithromycin (200 mg twice daily) as the first-line treatment. Medication adherence was confirmed through daily individual telephone calls with each participant.
Urea Breath Test (UBT) of H pylori eradication therapy | 8 weeks
  Success of the H pylori eradication was assessed 6 to 8 weeks after treatment using the urea breath test.

CONTACTS AND LOCATIONS:
Overall Officials: Yumiko Kamogawa, M.D., Ph.D., Study Director — NPO HIGAN
Locations (1):
- Khesar Gyalpo University of Medical Sciences of Bhutan, Thimphu, Thimphu District, Bhutan

IPD SHARING:
Plan to Share IPD: No